CLINICAL TRIAL: NCT06069362
Title: Prediction of Response to Manual Physiotherapy Using Somatosensory Profiles in Patients With Cervicobrachial Pain
Brief Title: Predictors of Response to Manual Physiotherapy Using Somatosensory Profiles in Patients With Cervicobrachial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Matia Foundation (Other); Osakidetza (Other)
Responsible Party: Principal Investigator, Xabat Casado, Physiotherapist, University of Deusto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FST_DCB
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cervical Radicular Pain; Cervical Radiculopathy; Cervical Pain
Keywords: Cervicobrachial pain; Nerve related neck arm pain
MeSH Terms: conditions — Radiculopathy; Neck Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual physiotherapy and neurodynamic exercises (Experimental): The treatment applied forms part of the routine clinical practice and includes the following:
  * Cervical passive mobilisation techniques and techniques of the anatomical structures surrounding the nerve root.
  * Home neurodynamic sliders of the upper limb and cervical mobility exercises.
  Interventions: Other: Manual physiotherapy and neurodynamic exercises

INTERVENTIONS:
Other: Manual physiotherapy and neurodynamic exercises — * Cervical passive mobilisation techniques and techniques of the anatomical structures surrounding the nerve. These techniques aim to open the nerve root foramen. They are gentle traction techniques and contralateral lateral glide mobilisation techniques. Interface techniques for scalenes will also be included.
  * Home exercises for cervical mobility and neurodynamic sliders of the upper extremity: Patients will be taught progressive upper extremity neurodynamic sliders, starting with gentle movement and progressing to exercises involving more movement based on the patient's irritability.
  Other Names: Manual physiotherapy and exercise

SUMMARY:
The goal of this clinical trial is to investigate about the characteristics that predict response to physiotherapy treatment in patients with nerve related neck arm pain. The main question to answer is whether there is a subgroup that responds better to physiotherapy treatment.

Participants will be assessed for clinical and neurophysiological characteristics prior to treatment. Afterwards they will receive 6 sessions of manual physiotherapy treatment along with home nerve gliding exercises once a week. Baseline measurements will be taken again after treatment to know if there have been any changes.

DETAILED DESCRIPTION:
During the first visit, socio-demographic data will be collected. Then, participants will be assessed using the quantitative sensory testing (QST) to evaluate the excitability of the nervous system. In addition, questionnaires and scales will be used to obtain information on the psychosocial factors involved, neuropathic pain characteristics and on the disability caused by their situation.

Finally, various clinical tests will be carried out to obtain information on neck movement and irritability at closure of the intervertebral foramen, mechanosensitivity of the upper limb with neurodynamic testing and alterations in sensitivity, strength and myotatic reflexes. Also they will be asked for permission to access to their imaging tests.

Once the pre-treatment data has been obtained, the manual physiotherapy and exercise treatment will begin, which aims to reduce the irritability of the nervous system.

Once the treatment is completed, the initial measurements will be repeated along with a global rating of change scale to classify patients as responders vs. non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with unilateral cervicobrachial pain

Exclusion Criteria:

* Signs of severe disease, cervical myelopathy, tumour, rheumatic diseases or a neurological pathology of central origin.
* Cervicobrachial pain of traumatic origin or as a result of whiplash.
* Previous surgical intervention of the cervical spine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Global rating of change scale | Pre-intervention and post-intervention at week 6 - Between intervention sessions, weekly. - Mid term: at week 14
  Is a self-administered questionnaire that aims to measure the degree of subjective improvement since the first intervention received. The questionnaire is scored with 7 positive items to assess the patient's subjective improvement progressively. It also presents 7 negative items to assess whether the patient has worsened. The 0 is defined as no improvement or worsening, the patient is the same.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Pre-intervention and post-intervention at week 6 - Mid term: at week 14
  Neck and arm pain over the last 24 hours will be assessed with the NPRS. 0 is considered as no pain and 10 as the worst pain imaginable.
Neck Disability Index | Pre-intervention and post-intervention at week 6 - Mid term: at week 14
  It is a unidimensional questionnaire consisting of 10 sections on different activities and measuring functionality.
Central Sensitization Inventory (CSI) | Pre-intervention and post-intervention at week 6
  CSI is a 25-item questionnaire to assess the presence of signs and symptoms consistent with central sensitisation.
Pain Detect Questionnaire (PD-Q) | Pre-intervention and post-intervention at week 6
  Questionnaire consisting of temporal and spatial pain descriptors and sensory descriptors. The PD-Q classifies patients into 3 groups as follows:
  * The result is negative = The neuropathic pain component is unlikely (Score 0 to 12).
  * The result is unclear = The result is ambiguous, however, the neuropathic pain component may be present (Score 13 to 18).
  * The result is positive = Neuropathic pain is likely to be present (Score 19 to 38).
  The intensity of the most intense and average pain during the last 4 weeks is recorded on an NPRS as part of the PD-Q.
Patient Specific Functional Scale (PSFS) | Pre-intervention and post-intervention at week 6
  PSFS is a scale that measures a patient's functional status by asking about activities that are difficult to perform based on their condition and scoring the level of limitation of each activity.
Tampa Scale of Kinesiophobia (TSK-11) | Pre-intervention and post-intervention at week 6
  It is an 11-item questionnaire developed to identify fear of of movement.
Patient Catastrophizing Scale | Pre-intervention and post-intervention at week 6
  It is a 13-item questionnaire developed to identify catastrophising thoughts or feelings in relation to painful experiences.
Scale for sleep quality | Pre-intervention and post-intervention at week 6
  An increasing scale of 0-10 will be used to assess the quality of sleep. 0 is considered to be very poor sleep quality as a result of the pain, and 10 is considered to be no sleep disturbance.
Hospital anxiety and depression scale | Pre-intervention and post-intervention at week 6
  Is one of the most widely used tests to measure anxiety and depression in a general population of patients.
Clinical examination | Pre-intervention and post-intervention at week 6
  The clinical examination will include a detailed anamnesis considering items published by other studies.
Sensitivity to touch | Pre-intervention and post-intervention at week 6
  The sensitivity to touch of the different dermatomes involved in the upper extremity will be evaluated by means of a piece of cotton and with a toothpick by means of the neuropen. The sensitivity of the healthy limb will be compared with that affected in upper extremity dermatomes. The patient should tell us if there are alterations in sensitivity and if he perceives the stimulus in a more noticeable, similar or lesser way. Results will be noted as hyperesthesia, normoestesia, or hypoesthesia.
Myotatic reflexes of the upper extremity | Pre-intervention and post-intervention at week 6
  The reflex hammer will be used to evaluate the response of the roots of C5 and C6 by percussion in the biceps tendon and percussion in the triceps tendon for the evaluation of the roots of C6 and C7. The healthy and affected limb will be examined and compared for asymmetries indicating pathology
Myotomes examination | Pre-intervention and post-intervention at week 6
  The loss of strength will be manually examined that would indicate a loss of function of different nerve roots.
Spurling test | Pre-intervention and post-intervention at week 6
  It consists of performing a homolateral inclination that aims to reduce the intervertebral foramen along with a compression. The test is considered positive with reproduction of symptoms.
Distraction test | Pre-intervention and post-intervention at week 6
  It consists of slightly pulling the cervical spine with the patient in supine position. The reduction of symptoms during the test is considered positive.
Extension + rotation test | Pre-intervention and post-intervention at week 6
  With the patient in supine position, an extension and homolateral rotation is performed. The reproduction of the symptoms suggests facet involvement in the patient's clinical picture.
Range of motion in rotation | Pre-intervention and post-intervention at week 6
  The patient will be asked to perform a bilateral active rotation. Limitation of mobility to the symptomatological ipsilateral side will be considered positive.
Examination of increased mechanosensitivity of nervous tissue | Pre-intervention and post-intervention at week 6
  It will be evaluated using neurodynamic tests of the upper extremity (ULNT1, ULNT 2 and ULNT 3) and palpation of the median, radial and ulnar nerves. ULNTs are passive brachial plexus and nerve provocation tests to be evaluated performed supine, involving a sequence of movements that gradually add tension to the nerve trunk. The test will be considered positive with reproduction of arm symptoms at least partially and with the presence of structural differentiation. Structural differentiation involves modifying some of the movements of the sequence away from the area of onset of symptoms. It is a feature frequently used to involve nerve tissue in the symptoms reproduced.
Pain mapping | Pre-intervention and post-intervention at week 6
  The participant will be asked to draw, on an electronic body map, the location and intensity of their symptoms.
Detection and thermal pain thresholds | Pre-intervention and post-intervention at week 6
  Part of the QST protocol standardised by the German Research Network on Neuropathic Pain will be applied.This includes detection and thermal pain thresholds.
  The thermal thresholds will be measured using the MSA Thermotest (Somedic) with 9 cm thermode. The reference temperature will be set at 32°C. The cutting temperatures will be 5ºC and 50ºC. All thresholds will be obtained with ramp stimuli (1ºC/sec) that will stop voluntarily when the subject presses a button. Firstly, the cold and heat detection thresholds will be evaluated, and finally the measurement of the cold and heat pain thresholds. The average threshold temperature of 3 valid consecutive measurements will be calculated for each parameter.
Vibration detection threshold | Pre-intervention and post-intervention at week 6
  It will be measured with a Rydel-Seiffer tuning fork (64 Hz, 8/8 scale). The threshold will be determined as a threshold of disappearance of perception with 3 repetitions of stimuli. Measurements will be taken over bony prominences unless the area of maximum pain does not exhibit a bony surface, in which case, measurements will be taken over adjacent soft tissue.
Pressure pain threshold | Pre-intervention and post-intervention at week 6
  It will be determined with a pressure algometer with a contact surface of 1 cm2 and a ramp speed of 50kPa/s (Somedic). Subjects will be asked to press a button when the sensation changes from pressure to pressure pain. The average value of the measurements in triplicate shall be used for the analysis.
Temporal summation of pain | Pre-intervention and post-intervention at week 6
  It will be measured by a repetitive pinprick stimulus at a controlled intensity using the set of pinprick stimulators (MRC systems). The perceived magnitude of a single puncture stimulus (256mN) will be compared to that of a series of 10 puncture stimuli of the same force repeated at a rate of 1/sec.
Conditioned pain modulation | Pre-intervention and post-intervention at week 6
  The cold pressor test will be used to evaluate the efficacy of endogenous pain inhibitory mechanisms. Patients will immerse the healthy limb's hand in an insulated container filled with cold water. The pressure pain threshold (PPT) test will be applied as a test stimulus to determine the potential effect of conditioned pain modulation during the application of the cold stimulus.
Offset Analgesia | Pre-intervention and post-intervention at week 6
  Using the thermode, we will identify the value for the heat pain threshold to obtain a value of 5/10 in the NPRS and then raise it by 1°C to obtain a new supra-threshold NPRS value. After a few seconds the temperature will be lowered back to the initial value and we will assess for changes in pain perception in the NPRS.
Magnetic resonance imaging and radiography | Pre-intervention
  The patient will be asked for permission to access the tests performed as part of the medical diagnosis, in order to study whether the morphological changes produced by the aging of the patient (baseline situation) can be predictors of the response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xabat Casado, PhD cand, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, San Sebastián, Gipuzkoa, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmid AB, Hailey L, Tampin B. Entrapment Neuropathies: Challenging Common Beliefs With Novel Evidence. J Orthop Sports Phys Ther. 2018 Feb;48(2):58-62. doi: 10.2519/jospt.2018.0603. PMID 29385943
- [Background] Bogduk N. On the definitions and physiology of back pain, referred pain, and radicular pain. Pain. 2009 Dec 15;147(1-3):17-9. doi: 10.1016/j.pain.2009.08.020. Epub 2009 Sep 16. No abstract available. PMID 19762151
- [Background] Vardeh D, Mannion RJ, Woolf CJ. Toward a Mechanism-Based Approach to Pain Diagnosis. J Pain. 2016 Sep;17(9 Suppl):T50-69. doi: 10.1016/j.jpain.2016.03.001. PMID 27586831

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT06069362/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT06069362/ICF_001.pdf